CLINICAL TRIAL: NCT03194373
Title: A Multi-Center Open Label Single Arm Phase II Trial Evaluating the Efficacy of Palbociclib in Combination With Carboplatin for the Treatment of Unresectable Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Trial Evaluating the Efficacy of Palbociclib in Combination With Carboplatin for the Treatment of Unresectable Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.054; HUM00130055 (Other: University of Michigan)
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — palbociclib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib and Carboplatin (Experimental): Treatment with Palbociclib and Carboplatin for up to 6 cycles:
  Palbociclib (Ibrance) (PO), dose= 125 mg PO daily, days=1-14, cycle length: 21 days Carboplatin (IV), dose= AUC 5, day= 1, cycle length: 21 days
  Maintenance Palbociclib after 6 cycles Palbociclib (Ibrance) 125 mg PO daily, days 1-21, cycle length: 28 days
  Interventions: Drug: Palbociclib; Drug: Carboplatin

INTERVENTIONS:
Drug: Palbociclib — Palbociclib (Ibrance) (PO), dose= 125 mg PO daily, days=1-14, cycle length: 21 days
  Maintenance Palbociclib:
  Palbociclib (Ibrance) 125 mg PO daily, days 1-21, cycle length: 28 days
Drug: Carboplatin — Carboplatin (IV), dose= AUC 5, day= 1, cycle length: 21 days

SUMMARY:
The purpose of this study is to test the effectiveness (how well the drug works), safety, and tolerability of the investigational drug combination of palbociclib (Ibrance) plus carboplatin in patients with metastatic head and neck squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented progressive squamous cell head and neck cancer with or without metastases, not amenable to curative treatment; or the patient has documented refusal of curative treatment.
* ECOG performance status of 0-2. Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.
* Presence of measurable disease by CT scan per RECIST v1.1.
* Age ≥18 years.
* Life expectancy of ≥12 weeks.
* Women of childbearing potential must have a negative serum or urine pregnancy test at time of screening and confirmed within 3 days prior to treatment. Women not of child-bearing potential will be defined as all women older than age 50 and anovulatory for 12 months.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Adequate organ and marrow function

Exclusion Criteria:

* Previous treatment with cytotoxic chemotherapy therapy in the recurrent/metastatic setting. Previous treatment with non-cytotoxic agents in the recurrent/metastatic setting is permitted. Gastrointestinal abnormalities causing impaired absorption precluding administration of oral medications.
* Evidence of untreated or progressive brain metastases, spinal cord compression, or carcinomatous meningitis.
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Patients (male and female) having procreative potential who are not willing or not able to use adequate contraception. Women who are pregnant or breast-feeding.
* Patients residing in prison.
* Prior experimental therapy within 30 days of enrollment.
* Availability of curative treatment option for the patient's cancer, whether surgery, chemotherapy, radiation, or combination thereof, unless the patient has documented refusal of curative treatment.
* Current use or anticipated inability to avoid use of drugs that are known strong CYP3A4/5 inhibitors (atazanavir, boceprevir, conivaptan, clarithromycin, grapefruit or grapefruit juice, indinavir, itraconazole, ketoconazole, nelfinavir, nefazodone, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole ).
* Current use or anticipated inability to avoid use of drugs that are known strong CYP3A4/5 inducers (carbamazepine, dexamethasone, fosphenytoin, phenytoin, phenobarbital, rifabutin, rifampin, rifapentine, St. John's wort).
* Patients with a history of severe allergic reaction to cisplatin or carboplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Swiecicki, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled patient withdrew prior to starting study treatment.
Groups:
- Palbociclib and Carboplatin: Treatment with Palbociclib and Carboplatin for up to 6 cycles: Palbociclib (Ibrance) 125 mg PO daily, days 1-14 + Carboplatin AUC 5 IV, day 1; cycle length 21 days.
  Maintenance Palbociclib after 6 cycles: Palbociclib (Ibrance) 125 mg PO daily, days 1-21; cycle length 28 days.
Period: Overall Study
Arm/Group | Palbociclib and Carboplatin
Started | 20
Received Palbociclib and Carboplatin (One participant received carboplatin but never received palbociclib) | 19
Completed (Evaluable for response) | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 21 patients enrolled; 18 were evaluable for response. One patient was not started on therapy after enrollment due to abrupt decline in performance status, another received carboplatin but never received palbociclib. A third patient was removed from study prior to imaging per physician discretion.
Arm/Group | Palbociclib and Carboplatin
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Number; unit: participants] — Population: 18 patients evaluable for response
  participants
    0 (Fully functional): number analyzed (Participants) | 18
    0 (Fully functional) | 8
    1 (Minor impairment): number analyzed (Participants) | 18
    1 (Minor impairment) | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Disease Control Rate (DCR)
Description: The primary clinical objective of this trial is to estimate disease control rate (DCR) at 12 weeks in patients with metastatic head and neck squamous cell cancer treated with carboplatin and palbociclib. DCR will be defined as either CR (Complete Response: Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.), PR (Partial Response: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.) or SD (Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.) at 12 weeks.
Time Frame: 12 weeks
Population: Patients were considered evaluable for response if they underwent response evaluation imaging after 2 cycles of receiving both carboplatin and palbociclib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib and Carboplatin
Number analyzed (Participants) | 18
percentage of participants | 33 [13 to 59]
Statistical Analysis 1: Comparison: Palbociclib and Carboplatin; Test type: Superiority — Power to detect a 20% improvement in disease control rate (DCR). Based on historical data, the DCR in R/M HNSCC with single agent platinum therapy is 40%. We hypothesize that addition of Palbociclib will increase DCR at 12 weeks to 60%. Two-stage design. Type I error rate of 0.059 and power of 0.80 when the true response rate is 0.60 with alpha=0.05. The two-stage sample size calculations assume a null probability of 0.40; Proportion = 33, 95% CI 2-sided [13 to 59]

2. Secondary Outcome: Median Progression Free Survival Time
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression. Progressive disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions. Estimated using a Kaplan-Meier analysis.
Time Frame: Up to 2 Years
Population: Patients were evaluable for survival if they underwent response evaluation imaging after 2 cycles of receiving both carboplatin and palbociclib.
Measure: Median (Full Range); unit: months
Arm/Group | Palbociclib and Carboplatin
Number analyzed (Participants) | 18
months | 2.9 [1.2 to 13.3]
Statistical Analysis 1: Comparison: Palbociclib and Carboplatin; Test type: Other; Median survival times were computed using the Kaplan-Meier method with standard error computed using Greenwood's formula. All analyses were done using SAS 9.4 software

3. Secondary Outcome: Median Overall Survival Time
Description: Overall survival is defined as the time from study enrollment to death from any cause. Estimated using a Kaplan-Meier analysis.
Time Frame: Up to 2 Years
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Palbociclib and Carboplatin
Number analyzed (Participants) | 18
months | 4.6 [1.4 to 14.8]
Statistical Analysis 1: Comparison: Palbociclib and Carboplatin; Test type: Other; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Treatment-related Toxicities
Description: Number of adverse events believed to be related (i.e., possibly, probably, or definitely) to palbociclib in combination with carboplatin, reported by grade according to the Common Terminology for Adverse Events version 4.0 (CTCAE v4).
Time Frame: Up to 2 years
Population: Patients were evaluable for treatment-related toxicities if they underwent response evaluation imaging after 2 cycles of receiving both carboplatin and palbociclib.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib and Carboplatin
Number analyzed (Participants) | 18
Participants
  Neutrophil count decreased : Grade 1-2 | 2
  Neutrophil count decreased : Grade 3-4 | 10
  Anemia : Grade 1-2 | 5
  Anemia : Grade 3-4 | 7
  White blood cell decreased : Grade 1-2 | 3
  White blood cell decreased : Grade 3-4 | 7
  Fatigue : Grade 1-2 | 7
  Fatigue : Grade 3-4 | 5
  Platelet count decreased : Grade 1-2 | 4
  Platelet count decreased : Grade 3-4 | 3
  Nausea : Grade 1-2 | 6
  Nausea : Grade 3-4 | 2
  Vomiting : Grade 1-2 | 2
  Vomiting : Grade 3-4 | 1
  Weight loss : Grade 1-2 | 4
  Weight loss : Grade 3-4 | 0
  Febrile neutropenia : Grade 1-2 | 0
  Febrile neutropenia : Grade 3-4 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment. All-cause mortality data was collected during entire study; 29 months.
Arm/Group | Palbociclib and Carboplatin
All-Cause Mortality (participants affected / at risk) | 16/19
Serious Adverse Events (participants affected / at risk) | 14/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib and Carboplatin (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Ataxia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - other (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Nervous system disorders - other (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib and Carboplatin (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 12 (28)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 12 (20)
Flu like symptoms (General disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lymphocyte count decreased (Investigations) | 6 (10)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 11 (19)
Pain (General disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 7 (15)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 10 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT03194373/Prot_SAP_000.pdf